

# Statistical Analysis Plan

Study: SC 2020-01

# STATISTICAL ANALYSIS PLAN

### Final v1.0

Protocol SC 2020-01 (Version 3.0, 02JUN2021)

Phase 1 Trial of IFx-Hu2.0 to Evaluate Safety in Patients with Skin Cancer

Date: October 26, 2021

### **TABLE OF CONTENTS**

| Tab | le of C | ontents | 2 |
|---|---|---|---|
| List | of Abb | previations | 4 |
| 1. | INTR | ODUCTION | 5 |
| 1 | .1 C | Objectives | 5 |
| | | Design | |
| 2. | Elabo | ration of Study Protocol | 5 |
| 2 | .1 S | Study Populations | 5 |
| 2 | .2 S | Study Endpoints | 5 |
| | 2.2.1 | Primary Endpoint | 5 |
| | 2.2.2 | Secondary Endpoints | 5 |
| | 2.2.3 | Exploratory Endpoint | 6 |
| 2 | .3 S | Sample Size | 6 |
| 3. | Statis | tical methods | 6 |
| 3 | | General | |
| 3 | .2 S | Subject Disposition, Demographics and Baseline Characters | 6 |
| | 3.2.1 | Safety Analysis | 6 |
| | 3.3.3. | Subgroup Analyses | 8 |
| 3 | | landling of Missing Data | |
| 3 | .5. P | Protocol Deviations | 8 |
| 3 | .6. Ir | nterim Analyses | 8 |
| 3 | .7. K | ey Data Items | 8 |
| | | Change to Planned Protocol Analysis | |
| 4. | OuTp | ut planned for the study report | 9 |
| 4 | .3. T | ables to be Included in Study Report | 9 |
| | 4.3.2. | | |
| | 4.3.3. | Demographic and Other Baseline Characteristics | 9 |
| | 4.3.4. | Summary of Safety Endpoints | 9 |
| 4 | .4. F | igures to be Included in the Clinical Study Report | 10 |
| 4 | .5. L | istings to be Included in the Clinical Study Report | 10 |
| | 4.5.2. | Listings of subject information | 10 |
| | 4.5.6. | Listings of safety data | 10 |
| 5. | | ences | |
| 6. | Attacl | nment: The Shells of Tables, Figures and Listings planned for Clinical Study Report | 11 |

#### **LIST OF ABBREVIATIONS**

**%RVT** Percent Residual Vial Tumor

AE Adverse Events

ANCOVA Analysis of Covariance
CI Confidence Interval

CTCAE Common Terminology Criteria for Adverse Events

DLT Dose Limiting Toxicity

DPS Data Presentation Specification
DSMB Data Safety Monitoring Board

ITT Intend-to-Treat

ICH International Committee for Harmonization

IP Investigational Product LSMEANS Least-squares Means

MedDRA Medical Dictionary for Drug Regulatory Affairs

PBRS Peachtree BioResearch Solution

PT Preferred Term

SAE Serious Adverse Events
SAP Statistical Analysis Plan
SAS Statistical Analysis System

SD Standard Deviation SOC System Organ Class

TEAE Treatment emergent adverse events

US United States

#### 1. INTRODUCTION

#### 1.1 Objectives

## **Primary Objective:**

· To assess safety and feasibility

#### **Secondary Objectives:**

• To assess post-therapeutic pathological response

#### **Exploratory Objectives:**

To assess anti-tumor immunity post-treatment.

### 1.2 Design

One hundred patients will receive IFx-Hu2.0 on an outpatient basis at a single time point in a single lesion. These patients will be assessed for any immediate adverse reactions and at Week 4 (Day 28+/-5 days) for any delayed adverse events.

#### 2. ELABORATION OF STUDY PROTOCOL

### 2.1 Study Populations

 Safety Analysis Dataset: the subset of participants who received at least one dose of study intervention (IFx-Hu2.0). All safety analyses will be conducted on Safety Analysis Set.

#### 2.2 Study Endpoints

#### 2.2.1 Primary Endpoint

The primary endpoints of this trial will be the safety and feasibility of the treatment regimen. Safety will be reported using the most current version of the Common Terminology Criteria for Adverse Events (CTCAE).

Feasibility will be defined as the ability to treat at least 85 of the approximate 100 patients enrolled without investigational product (IP) related dose-limiting toxicity (DLT).

A DLT is defined as an adverse event equal to or greater than grade 3, at least possibly related to the investigational agent, occurring within a 4-week period following IP administration.

#### 2.2.2 Secondary Endpoints

The secondary endpoint is Pathological Response defined as a response assessment to IFx-Hu2.0 in tumor lesions excised by evaluating percent Residual Vial Tumor (%RVT), at four weeks as:

- Pathological complete response (pCR),
- Major pathological response (mPR),
- Partial pathological response (pPR), or

Pathological non-response (pNR))

#### 2.2.3 Exploratory Endpoint

Patient samples (plasma and/or serum) will be assayed to detect tumor antigen specific antibody generation in addition to a protein biomarker discovery assay specific to immuno-oncology therapy assessments.

IHC will be performed on pre- and post-treatment tissue samples to contrast the cell sub-types across time points.

# 2.3 **Sample Size**

The intent of this study is to enroll approximately 100 evaluable patients to assess the safety of IFx-Hu2.0 as a monotherapy. A sample size of 100 has the following precision for estimation of DLT rates ranging from 0.1 to 0.5. A DLT is defined as an adverse event equal to or greater than grade 3, at least possibly related to the investigational agent, occurring within a 4-week period following IP administration, and deemed as having unacceptable toxicity by the principal investigator and/or medical monitor. Precision is measured by 1-sided 95% upper confidence limit on the estimated DLT rate via exact binomial distribution. For example, if no DLT is observed in patients on IFX-Hu 2.0, then the true underlying DLT rate is lower than 0.099 with 95% confidence.

#### 3. STATISTICAL METHODS

#### 3.1 General

All data will be analyzed using the Statistical Analysis System (SAS®; Version 9.2 or higher). Continuous variables will be summarized using descriptive statistics, including sample size, mean, standard deviation (SD), median, minimum, and maximum. Categorical variables will be summarized using number and percent of subjects for each outcome.

All statistical tests will be two sided, and statistical significance level is 0.05.

#### 3.2 Subject Disposition, Demographics and Baseline Characters

- Reasons for withdrawal will be summarized.
- Demographics and baseline characters will be summarized on safety analysis set using descriptive statistics.
- Medical history will be summarized with MedDRA system organ class (SOC) and preferred term (PT) for Safety analysis set.
- Prior and concomitant medications will be summarized with WHO Drug Class 3 name for Analysis of Study Endpoints

#### 3.2.1 Safety Analysis

The safety analysis will be conducted on safety analysis set that includes all treated subjects.

Safety endpoints will be analyzed as summary statistics during treatment and/or as change scores from baselines such as shift tables. Treatment emergent adverse events (TEAEs) will be coded using Medical Dictionary for Regulatory Activities (MedDRA). TEAE severity and relationship to study treatment will be presented by dose cohort, MedDRA system organ class (SOC) and preferred term (PT).

The information reported about each AE will be the start date, stop date, severity, relationship, outcome, and duration). AEs leading to premature discontinuation from the study and serious treatment emergent AEs will be presented with either a summary table or a data listing.

#### Adverse Events

TEAEs are defined as signs or symptoms that emerge during treatment or within 28 days of the last dose of Investigational Product, including those signs and symptoms that have been absent pre-treatment or that have worsened relative to the pre-treatment assessment. Any adverse event considered related to treatment will also be considered a TEAE, regardless of the elapsed time since the last dose of Investigational Product.

Number and percentage of subject with any DLT will be reported by dose cohort, MedDRA SOC and PT. Overall DLT rate for safety analysis set will be provided with 95%CI.

Number and percentage of subject with any TEAEs will be summarized by MedDRA SOC, PT, intensity, and relationship to the study treatment.

Number and percentage of subject with serious TEAE will also be summarized and listed.

#### Vital Signs

The observed vital signs at each visit and the change from baseline to each post-baseline visit will be summarized by cohort using descriptive statistics.

#### Physical Examination

Abnormal findings in the physical examination will be summarized by dose cohort using descriptive statistics.

#### Clinical Laboratory Tests

Clinical laboratory test values outside the normal range and clinically significant abnormal range will be flagged in the data listing. Laboratory data will be summarized by cohort using shift tables (baseline to notable post-baseline visit). The change from baseline will be summarized using descriptive statistics.

#### ECOG

The data observed from ECOG performance status will be summarized appropriately.

#### • ECG

The results of ECGs will be summarized appropriately.

#### 3.3.2. Exploratory Analyses

Patient samples (plasma and/or serum) will be assayed to detect tumor antigen specific antibody generation in addition to a protein biomarker discovery assay specific to immuno-oncology therapy assessments.

# 3.3.3. Subgroup Analyses

No subgroup analyses of safety endpoints will be planned.

### 3.4. Handling of Missing Data

Missing data will not be imputed for safety analyses.

#### 3.5. Protocol Deviations

Listing for all protocol deviations will be provided.

### 3.6. Interim Analyses

Interim analysis will not be planned.

# 3.7. Key Data Items

### **Study Analysis Population Definition:**

Safety analysis set: All enrolled patients who have received at least 1 dose of IFx-Hu2.0.

#### **Important Derived Variables:**

- Age = (Screening Date Date of Birth +1)/365.25.
- Prior Medications and Treatments: the medications and treatments started before enrolled to the study.
- Concomitant Medication and Treatments: the medications and treatments started after being enrolled to the study.
- Baseline: Day 0 (Baseline Visit). All clinical measurements collected at Day 0 or before the dose of IFx-Hu2.0 on Day 0 will be analyzed as baseline.
- Post Baseline (post dose): All clinical measurements collected after the dose of IFx-Hu2.0 on Day 0 will be analyzed as post baseline.
- Dose-Limiting Toxicity (DLT): Treatment emergent adverse event (TEAE) equal to or greater than grade 3, at least possibly related to the investigational agent, occurring within a 4-week period following IFx-Hu2.0 administration

#### 3.8. Change to Planned Protocol Analysis

Not applicable.

#### 4. OUTPUT PLANNED FOR THE STUDY REPORT

### 4.3. Tables to be Included in Study Report

In the following sections, the different results are presented in the order in which it is planned to make them appear in the study report.

The table templates are available in the Appendix of the SAP. The content shown in the templates is only meant as an example. It is not based on real study data or details concerning design.

#### 4.3.2. Summary of Subject Information

Table 14.1.1.1 Subject Disposition – Safety Analysis Set

# 4.3.3. Demographic and Other Baseline Characteristics

- Table 14.1.2.1 Summary of Demographics Safety analysis set
- Table 14.1.2.2 Number (%) of Subjects with Medical History by MedDRA System Organ Class and Preferred Term Safety Analysis Set
- Table 14.1.2.3 Number (%) of Subjects with Current Medical Conditions by MedDRA System Organ Class and Preferred Term Safety Analysis Set
- Table 14.1.2.4 Number (%) of Subjects with Prior Medications by WHO Drug Class 3 Name and Preferred Term Safety Analysis Set
- Table 14.1.2.5 Number (%) of Subjects with Concomitant Medications by WHO Drug Class 3
  Name and Preferred Term Safety Analysis Set

#### 4.3.4. Summary of Safety Endpoints

- Table 14.3.1.1 Overall Summary of Adverse Events Safety Analysis Set
- Table 14.3.1.2 Number (%) of Subjects with TEAEs by SOC and PT Safety Analysis Set
- Table 14.3.1.3 Number (%) of Subjects with DLT by MedDRA SOC and PT Safety Analysis Set
- Table 14.3.1.4 Number (%) of Subjects with Serious TEAE by MedDRA SOC and PT Safety Analysis Set
- Table 14.3.1.5 Number (%) of Subjects with Study Treatment Related TEAE by MedDRA SOC and PT Safety Analysis Set
- Table 14.3.1.6 Number (%) of Subjects with Immune Response Treatment Emergent Adverse Events Safety Analysis Set
- Table 14.3.1.7 Number (%) of Subjects with TEAE by MedDRA Preferred Term and Overall Frequency Safety Analysis Set
- Table 14.3.2.1Summary of Chemistry Laboratory Tests by Visit Safety Analysis Set
- Table 14.3.2.2 Summary of Hematology Laboratory Tests by Visit Safety Analysis Set
- Table 14.3.2.3 Summary of Urinalysis Laboratory Tests by Visit Safety Analysis Set
- Table 14.3.2.4 Summary of Qualitative Urinalysis Laboratory Tests by Visit Safety Analysis Set
- Table 14.3.2.5 Shift Tables of Laboratory Results from Baseline to the Worst Post-Baseline Visit (Chemistry) Safety Analysis Set
- Table 14.3.2.6 Shift Tables of Laboratory Results from Baseline to the End of Study (Chemistry) Safety Analysis Set

- Table 14.3.2.7 Shift Tables of Laboratory Results from Baseline to the Worst Post-Baseline Visit (Hematology) Safety Analysis Set
- Table 14.3.2.8 Shift Tables of Laboratory Results from Baseline to the End of Study (Hematology) Safety Analysis Set
- Table 14.3.2.9 Shift Tables of Laboratory Results from Baseline to the Worst Post-Baseline Visit (Urinalysis) Safety Analysis Set
- Table 14.3.2.10 Shift Tables of Laboratory Results from Baseline to the End of Study (Urinalysis) Safety Analysis Set
- Table 14.3.3.1 Summary of Vital Signs and Change from Baseline Safety Analysis Set
- Table 14.3.4.1 Number (%) of Subject with Abnormal Physical Examinations Safety Analysis Set
- Table 14.3.5.1 Number (%) of Subject with ECOG Performance Status Safety Analysis Set
- Table 14.3.6.1 Number (%) of Subject with Abnormal ECG Safety Analysis Set
- Table 14.3.7.1 Summary of Pathological Response Safety Analysis Set

#### 4.4. Figures to be Included in the Clinical Study Report

No figures are planned for this study.

#### 4.5. Listings to be Included in the Clinical Study Report

#### 4.5.2. Listings of subject information

- Listing 16.2.1.1 Subject Disposition Safety Analysis Set
- Listing 16.2.2.1 Protocol Deviations Safety Analysis Set

#### 4.5.3. Demographics and Baseline Characters

- Listing 16.2.4.1 Demographic and Baseline Characteristics Safety Analysis Set
- Listing 16.2.4.2 Subjects with Past and Current Medical Conditions Safety Analysis Set
- Listing 16.2.4.3 Subjects with Prior Medications Safety Analysis Set
- Listing 16.2.4.4 Subjects with Concomitant Medications Safety Analysis Set
- Listing 16.2.4.5 Subjects with Disease Characteristics for Primary Tumor Type Safety Analysis Set

#### 4.5.4. Study Drug Exposure

Listing 16.2.5.1 Study Drug Exposure – Safety Analysis Set

#### 4.5.5. Lesion Evaluation

Listing 16.2.6.1 Injected Lesion Evaluation – Safety Analysis Set

#### 4.5.6. Listings of safety data

- Listing 16.2.7.1 Treatment Emergent Adverse Events Safety Analysis Set
- Listing 16.2.7.2 Serious Treatment Emergent Adverse Events Safety Analysis Set
- Listing 16.2.7.3 Treatment Emergent Adverse Events of DLT Safety Analysis Set
- Listing 16.2.7.4 Study Treatment Related Adverse Events Safety Analysis Set

Listing 16.2.7.5 Immune Response Treatment Emergent Adverse Events – Safety Analysis Set

Listing 16.2.7.6 Treatment Emergent Adverse Events Leading to Study Discontinuation - Safety Analysis Set

Listing 16.2.8.1 Chemistry Laboratory Tests - Safety Analysis Set

Listing 16.2.8.2 Hematology Laboratory Tests - Safety Analysis Set

Listing 16.2.8.3 Urinalysis Laboratory Tests - Safety Analysis Set

Listing 16.2.8.4 Pregnancy Tests - Safety Analysis Set

Listing 16.2.9.1 Vital Signs - Safety Analysis Set

Listing 16.2.9.2 12-Lead Electrocardiograms - Safety Analysis Set

Listing 16.2.9.3 ECOG Performance Status - Safety Analysis Set

Listing 16.2.9.4 Physical Examinations - Safety Analysis Set

Listing 16.2.10.1 Pathological Response Results - Safety Analysis Set

| _ | _ | <br>, | $\sim$ |
|----------|--------------------|---------------|--------|
| <b>h</b> | $\boldsymbol{\nu}$ | , <b>–</b> NI | CFS |

Protocol: Phase 1 Trial of IFx-Hu2.0 to Evaluate Safety in Patients with Skin Cancer, Version 3.0, 02 Jun 2021, Morphogenesis, Inc.

6. ATTACHMENT: THE SHELLS OF TABLES, FIGURES AND LISTINGS PLANNED FOR CLINICAL STUDY REPORT



# Statistical Analysis Plan

Study: SC 2020-01

# Approval for Statistical Analysis Plan

Title: Phase 1 Trial of IFx-Hu2.0 to Evaluate Safety in Patients with Skin

Cancer

Reference: SC 2020-01/SAP

Version: 1.0

Date effective:

Author: Dion Chen PhD., Peachtree BRS

Author's signature: Sion Chen Date: 10/27/2021

The above Statistical Analysis Plan has been reviewed and approved by the Sponsor:

Name of **Ashraf Dehlawi** 

Reviewer/Approver

Position: Sr. Director of Development Operations, Morphogenesis, Inc.

Signature for

sponsor: Oshraf Dehlawi Date: 10/28/2021

# RightSignature

# SIGNATURE CERTIFICATE



#### REFERENCE NUMBER

502B6A0B-41AD-4D35-865E-109EBBE008AA

#### **DOCUMENT DETAILS** TRANSACTION DETAILS

**Reference Number** 

502B6A0B-41AD-4D35-865E-109EBBE008AA

**Transaction Type** 

Signature Request

Sent At

10/27/2021 18:27 EDT

**Executed At** 

10/28/2021 09:22 EDT

**Identity Method** 

**Distribution Method** 

email

Signed Checksum

e8ae 506 ed ca 88 d0 61 da 6cc e9ac 31 be 3f0 e3e16c0 bb 4b8f26195cf be 3d9f9a28a

**Signer Sequencing** 

Disabled

**Document Passcode** 

Disabled

**Document Name** 

Sc 2020-01 Sap Final V1 0 26oct2021

**Filename** 

 $sc\_2020\text{-}01\_sap\_final\_v1\_0\_26oct2021.docx$ 

**Pages** 

12 pages

**Content Type** 

application/vnd.openxmlformats-officedocument.wordprocessingml.document

File Size 96.5 KB

**Original Checksum** 

 $\tt d68d2164c47a51c9714b9507c26b134d74d4a2e4b62fe32b4ebfe80c7c913d8d$ 

# SIGNERS

| SIGNER | E-SIGNATURE | EVENTS |
|---|---|---|
| Name<br>Ashraf Dehlawi | <b>Status</b> signed | Viewed At<br>10/28/2021 09:22 EDT |
| Email adehlawi@morphogenesis-inc.com Components 2 | Multi-factor Digital Fingerprint Checksum Obfdd6e955adfdf816cc185b7d5d82e011caadafe0ec41a34945f196f3c265a9 IP Address 47.206.102.135 Device Chrome via Windows Typed Signature | Identity Authenticated At<br>10/28/2021 09:22 EDT<br>Signed At<br>10/28/2021 09:22 EDT |
| | Oshraf Behlawi Signature Reference ID 4E4B4069 | |

#### Name Dion Chen

# **Email**

dion.chen@peachtreebrs.com

#### Components

# Status

signed

# **Multi-factor Digital Fingerprint Checksum**

7509ba757c1013e722c1d61ccba3eff5decbce821e56247d7c1cc6ddbbbd9e5a

#### **IP Address**

74.103.183.55

#### Device

Chrome via Windows

#### Typed Signature

Bion Chen

#### Signature Reference ID

88FA280A

# Viewed At

10/27/2021 20:14 EDT

# **Identity Authenticated At**

10/27/2021 20:15 EDT

#### Signed At

10/27/2021 20:15 EDT

# **AUDITS**

| TIMESTAMP | AUDIT |
|---|---|
| 10/27/2021 18:27 EDT | Sara Moore (sara.moore@peachtreebrs.com) created document 'sc_2020-01_sap_final_v1_0_26oct2021.docx' on Chrome via Windows from 71.229.81.117. |
| 10/27/2021 18:27 EDT | Dion Chen (dion.chen@peachtreebrs.com) was emailed a link to sign. |
| 10/27/2021 18:27 EDT | Ashraf Dehlawi (adehlawi@morphogenesis-inc.com) was emailed a link to sign. |
| 10/27/2021 18:28 EDT | Ashraf Dehlawi (adehlawi@morphogenesis-inc.com) was emailed a reminder. |
| 10/27/2021 18:28 EDT | Dion Chen (dion.chen@peachtreebrs.com) was emailed a reminder. |
| 10/27/2021 20:14 EDT | Dion Chen (dion.chen@peachtreebrs.com) viewed the document on Chrome via Windows from 74.103.183.55. |
| 10/27/2021 20:15 EDT | Dion Chen (dion.chen@peachtreebrs.com) authenticated via email on Chrome via Windows from 74.103.183.55. |
| 10/27/2021 20:15 EDT | Dion Chen (dion.chen@peachtreebrs.com) signed the document on Chrome via Windows from 74.103.183.55. |
| 10/28/2021 09:22 EDT | Ashraf Dehlawi (adehlawi@morphogenesis-inc.com) viewed the document on Chrome via Windows from 47.206.102.135. |
| 10/28/2021 09:22 EDT | Ashraf Dehlawi (adehlawi@morphogenesis-inc.com) authenticated via email on Chrome via Windows from 47.206.102.135. |
| 10/28/2021 09:22 EDT | Ashraf Dehlawi (adehlawi@morphogenesis-inc.com) signed the document on Chrome via Windows from 47.206.102.135. |